CLINICAL TRIAL: NCT00303901
Title: Percutaneous Thoracic Cryotherapy (PTC) for Inoperable Primary Lung Cancer and Metastatic Management
Brief Title: Cryotherapy in Treating Patients With Primary Lung Cancer or Lung Metastases That Cannot Be Removed By Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Peter John Littrup, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000462091; P30CA022453 (NIH); WSU-C-2975; WSU-0509002942
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Lung Cancer; Metastatic Cancer
Keywords: lung metastases; recurrent non-small cell lung cancer; recurrent small cell lung cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; extensive stage small cell lung cancer; limited stage small cell lung cancer; pulmonary carcinoid tumor
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Cryosurgery; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cryosurgery (Experimental): cryoprobe is placed in the proper position using CT imaging guidance, and as internal tissue is being frozen, the physician avoids damaging healthy tissue by viewing the movement of the probe on CT images transmitted to a monitor similar to a television screen. Living tissue, healthy or diseased, cannot withstand extremely cold conditions.
  Interventions: Procedure: cryosurgery; Procedure: positron emission tomography

INTERVENTIONS:
Procedure: cryosurgery
Procedure: positron emission tomography

SUMMARY:
RATIONALE: Cryotherapy kills tumor cells by freezing them. This may be an effective treatment for primary lung cancer or lung metastases that cannot be removed by surgery.

PURPOSE: This clinical trial is studying how well cryotherapy works in treating patients with primary lung cancer or lung metastases that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Estimate the local and distant failure rates after percutaneous thoracic cryotherapy (PTC) in patients with unresectable primary lung cancer or lung metastases.
* Estimate rates of PTC complications and adverse reactions.
* Determine the correlations between procedural parameters and follow-up imaging parameters, with the latter being used as surrogates of local and/or distant treatment failure.

OUTLINE: Patients undergo CT-guided percutaneous thoracic cryotherapy over 2 hours under local or general anesthesia. Grouped cryoprobes are inserted into the tumor, utilizing a freeze-thaw-freeze cycle, creating cytotoxic temperatures (less than -20°C to -40°C) that encompass the entire anticipated tumor volume.

Patients undergo positron emission tomography at baseline and after cryotherapy to assess tumor standard uptake variable.

After completion of study treatment, patients are followed at 1, 3, 6 and 12 months.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed malignant pulmonary neoplasm
* New lung lesion(s) with definitive clinical and imaging features of primary or metastatic disease allowed

  * Imaging findings compatible with localized treatment failure after prior cryotherapy allowed
* Malignant pleural effusion allowed provided it is associated with a distinct measurable pulmonary mass amenable to cryotherapy
* Metastatic disease must meet all of the following criteria:

  * Primary tumors have been resected or have been deemed controlled by other therapies
  * No other widespread metastases evident (e.g., multiple hepatic or brain metastases)
* Each pulmonary mass must be amenable to CT-guided percutaneous cryotherapy approach
* No more than 5 targeted masses for study therapy

  * Target mass defined as pulmonary, hilar, mediastinal, and/or chest wall mass > 1 cm, but < 10 cm in average diameter
* Unresectable disease by surgical consultation OR patient refused surgical options
* Nonenhanced and enhanced CT scan required within the past 6 weeks done at 4-5 mm increments with available soft tissue and mediastinal windows to assess size and extent of all thoracic tumors

  * PET scan required within the past 6 months noting the correlation with the above CT locations, if not already obtained by a combined PET/CT scanner

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) > 60-100% OR WHO/ECOG/Zubrod PS 0-2
* FEV_1 > 30% of predicted
* DLCO > 40% of predicted
* Platelet count ≥ 70,000/mm^3
* INR < 1.5
* No uncontrolled coagulopathy or bleeding diathesis
* Not pregnant or nursing
* Negative pregnancy test
* No serious medical illness, including any of the following:

  * Uncontrolled congestive heart failure
  * Uncontrolled angina
  * Myocardial infarction
  * Cerebrovascular event within 6 months prior to study entry
* No medical contraindication or potential problem that would preclude study compliance

PRIOR CONCURRENT THERAPY:

* At least 7 days since prior aspirin and aspirin-like medications
* At least 3 days since prior warfarin, clopidogrel bisulfate, or similar compounds
* No concurrent drugs causing bleeding tendencies (e.g., aspirin, warfarin, or clopidogrel bisulfate)
* No concurrent participation in other experimental studies

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Littrup, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cryosurgery: cryoprobe is placed in the proper position using CT imaging guidance, and as internal tissue is being frozen, the physician avoids damaging healthy tissue by viewing the movement of the probe on CT images transmitted to a monitor similar to a television screen. Living tissue, healthy or diseased, cannot withstand extremely cold conditions.
  cryosurgery
  positron emission tomography
Period: Overall Study
Arm/Group | Cryosurgery
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cryosurgery
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Local Failure Rates by CT Scan
Description: Local Failure Rates by CT Scan Assessed as Percentage of Participants with Local Recurrence
Time Frame: at 3, 6, and 12 months
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | Cryosurgery
Number analyzed (Participants) | 40
% of participants | 15 [7 to 29]

2. Primary Outcome: Distant Failure Rate
Description: Distant Failure Rates by CT Scan Assessed as Percentage of Participants with Local Recurrence
Time Frame: at 3, 6, and 12 months
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | Cryosurgery
Number analyzed (Participants) | 40
% of participants | 52.5 [37 to 67]

3. Secondary Outcome: Rate of Complications and Adverse Reactions by Occurrences of Toxicities
Description: Rate of complications and adverse reactions by occurrences of toxicities as measured by the number of participants with a given category of toxicity.
Time Frame: at 3, 6, and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cryosurgery
Number analyzed (Participants) | 40
Participants
  DVT | 1
  atelectasis | 3
  constipation | 2
  contact dermatitis | 1
  deconditioning | 1
  depression | 1
  epigastric pain | 1
  fatigue | 3
  hemothorax | 1
  insomnia | 1
  muscle spasm | 1
  pain right side | 1
  severe atrial flutter | 1
  Anemia | 7
  Chest Wall Pain | 21
  Cough | 6
  Dyspnea | 7
  Elevated AST | 1
  Hemoptysis | 8
  Hemorrhagic Effusion | 1
  Hypotension | 1
  Hypoxia | 2
  Pleural Effusion | 21
  Pneumothorax | 21
  Pulmonary Hemorrhage | 16
  anxiety | 1
  blister | 1
  blurriness of vision | 1
  bradycardia | 1
  cardiac arrest | 1
  elevated ALT | 1
  headache | 1
  heartburn/dyspepsia | 1
  hepatic arteriovenous fistula | 1
  hyperglycemia | 1
  hypertension | 1
  ileus | 1
  infection | 1
  infection with normal ANC | 1
  low phosphorous | 1
  lymphopenia | 3
  nausea | 2
  pain | 1
  pneumonitis | 1
  progressive weakness | 1
  respiratory failure | 1
  subcutaneous hematoma | 1
  thrombocytopenia | 1
  vomiting | 2

4. Secondary Outcome: Correlate Procedural Parameters and Follow-up Imaging Parameters
Time Frame: at 3, 6, and 12 months
Reporting Status: Not Posted

5. Secondary Outcome: Point and Exact Confidence Interval Estimates of Patients Who Undergo Multiple Cryotherapy Procedures
Time Frame: 12 months after the last patient was enrolled
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Cryosurgery
Serious Adverse Events (participants affected / at risk) | 9/40
Other Adverse Events (participants affected / at risk) | 38/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cryosurgery (N=40)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Hepatic arteriovenous fistua (Renal and urinary disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Infection with normal ANC (Infections and infestations) | 1 (1)
Progressive weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Deep vein thrombosis (DVT) (Vascular disorders) | 1 (1)
Deconditioning (General disorders) | 1 (1)
Severe atrial flutter (Cardiac disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cryosurgery (N=40)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 7 (7)
Chest wall pain (Cardiac disorders) | 21 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 21 (21)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 21 (21)
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 16 (16)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
There were no study limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No